CLINICAL TRIAL: NCT01581736
Title: Molecular Regulation of Muscle Glucose Metabolism
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI job change
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Lori R. Roust, Consultant in Endocrinology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-004005
Record Dates: First submitted 2012-02-15; First posted 2012-04-20 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: insulin resistance; mitochondria
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin, Regular, Human; Insulin; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): Proteomics of muscle after a single bout of exercise compared to baseline with U100 Humulin infusion at rate of 80 milliunits(mU)/m^2 surface area.
  Interventions: Drug: U100 Humulin; Other: Exercise

INTERVENTIONS:
Drug: U100 Humulin — Infused at a rate of 80/mU/m2 surface area per minute one time over 2 hours
  Other Names: Humulin; Human insulin
Other: Exercise — Single episode of exercise riding a stationary bike.

SUMMARY:
This protocol is being conducted to determine the mechanisms responsible for insulin resistance, obesity and type 2 diabetes.

DETAILED DESCRIPTION:
This protocol involves performance of a hyperinsulinemic euglycemic clamp with 2 muscle biopsies and an exercise study with a muscle biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
2. Subjects may be of either sex, age as described in each protocol. Female subjects must be non-lactating and must either be at least two years post-menopausal, (if diabetic or obese) or be using adequate contraceptive precautions (i.e. oral contraceptives, approved hormonal implant, intrauterine device, diaphragm with spermicide, condom with spermicide), or be surgically sterilized (i.e. bilateral tubal ligation, bilateral oophorectomy). Female patients (except for those patients who have undergone a hysterectomy or bilateral oophorectomy) are eligible only if they have a negative pregnancy test throughout the study period.
3. Subjects must range in age as described in each specific protocol.
4. All nondiabetic subjects must have normal oral glucose tolerance.
5. Subjects must have the following laboratory values:

   1. Hematocrit ≥ 35 vol%
   2. Serum creatinine ≤ 1.6 mg/dl
   3. Aspartate aminotransferase (AST) (SGOT) < 2 times upper limit of normal
   4. Alanine aminotransferase (ALT) (SGPT) < 2 times upper limit of normal
   5. Alkaline phosphatase < 2 times upper limit of normal
   6. Triglycerides < 150 mg/dl.
   7. Prothrombin time (PT) 11.7 -14.3 (During Liposyn/heparin infusion, PT will be determined to insure that it is < 1.5-2.0 times the normal value.)
   8. Partial thromboplastin time (PTT) 23.0-37.0.

Exclusion Criteria:

1. Subjects must not be receiving any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on stable dose of such agents for the past three months before entry into the study. Subjects may be taking a stable dose of estrogens or other hormonal replacement therapy, if the subject has been on these agents for the prior three months. Subjects taking systemic glucocorticoids are excluded.
2. Subjects with a history of clinically significant heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the EKG), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) will not be studied.
3. Recent systemic or pulmonary embolus, untreated high-risk proliferative retinopathy, recent retinal hemorrhage, uncontrolled hypertension, systolic BP > 180, diastolic BP > 105, autonomic neuropathy, resting heart rate > 100, electrolyte abnormalities.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | one month from date of volunteer study
  euglycemic clamp

SECONDARY OUTCOMES:
acetylation of mitochondrial adenine nucleotide translocase | within 6 months of volunteer study
  proteomics analysis of post translational modification of proteins obtained from isolated mitochondria

CONTACTS AND LOCATIONS:
Overall Officials: Lori Roust, MD, Principal Investigator — Mayo Clinic; Lawrence J. Mandarino, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States